CLINICAL TRIAL: NCT04507971
Title: Effects of MET-3 and MET-5 on Gut Microbiome and Metabolic Function in Men and Women With Hypertriglyceridemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: NuBiyota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MET-5 101
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Obesity, Metabolically Benign
MeSH Terms: conditions — Obesity, Metabolically Benign

STUDY DESIGN:
Intervention Model Description: There are two parallel treatment arms. Responders to either treatment will continue with their assigned treatment through to the end of the study. Non-responders will cross-over to the other treatment at week 4 of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MET-3 2.5 g daily for 4 weeks (Experimental): MET-3 is composed of twenty-two strains of bacteria and was designed to treat metabolic syndrome. The strains that were selected are based on strains that are known butyrate producers, associated with healthy subjects and improved gut barrier function. MET-3 is provided in capsule form and 5 capsules will be swallowed by each subject once daily for 4 weeks.
  Interventions: Biological: MET-3
- MET-5 2.5 g daily for 4 weeks (Experimental): MET-5 is a new product composed of twenty-six strains of bacteria isolated from the stool of a different healthy donor than MET-3. Although it is expected to work in a similar fashion to MET-3, it contains some strains that are unique in comparison to the original MET-3 formulation and have been associated with leanness in the scientific literature. MET-5 is provided in capsule form and 5 capsules will be swallowed by each subject once daily for 4 weeks.
  Interventions: Biological: MET-3

INTERVENTIONS:
Biological: MET-3 — Human microbiome supplementation derived from bacterial strains isolated from fecal matter and grown in a laboratory environment
  Other Names: MET-5

SUMMARY:
The purpose of this pilot study is to determine the effects of two human microbiome formulations (MET-3 and MET-5) on fasting serum TG concentration.

DETAILED DESCRIPTION:
Obesity is a condition characterized by an excess amount of body fat, and is defined as a body mass index (BMI) of 30 kg/m² or greater. The rising prevalence of obesity in all parts of the world is of great public health concern due to the fact that obesity is associated with many causes of morbidity and mortality. Excess body fat accumulates when energy intake is greater than energy expenditure and recently, the role of the colonic microbiome has been highlighted as a potential contributor to energy balance. The obese microbiome is suggested to promote obesity due to an excess production of short-chain fatty acids, and, thus, increased colonic energy availability.

The purpose of this pilot study is to determine the effects of two human microbiome formulations (MET-3 and MET-5) on fasting serum TG concentration.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating females who are taking adequate contraceptive precaution, aged 18 to 49 years inclusive;
2. Body Mass Index (BMI) ≥25.0 kg/m2 and ≤40.0 kg/m2;
3. Stable body weight (±4 kg) for the past 4 months with no intention to gain or lose weight;
4. Fasting serum triglycerides ≥1.5 mmol/L (133 mg/dL) and <8 mmol/L (<709 mg/dL) at screening;
5. Fasting serum glucose <7.0 mmol/L (<126 mg/dl);
6. HbA1c <6.5% at screening;
7. Blood pressure <160/100;
8. AST, ALT and ALP ≤3 times the upper limit of normal (liver function) at screening;
9. Serum creatinine < 1.5 times the upper limit of normal (kidney function) at screening;
10. Willing to maintain habitual diet, physical activity pattern, and body weight throughout the trial;
11. Willing to refrain from taking probiotic supplements throughout the trial;
12. Willing to abstain from strenuous exercise, consuming alcoholic drinks 24 hours before study days and during study days;
13. Willing to maintain current dietary supplement and medication use throughout the trial. On test days, subject agrees to bring any dietary supplements or medications taken in the morning with them to the clinical site to take just prior to the glucose test meal;
14. Subject is not currently participating nor recently (within 30 days of screening) participated in a clinical trial involving long-term exposure (greater than 24 hours) to an investigational drug, nutritional supplement or lifestyle modification;
15. Understanding the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study investigator and other authorized agents as indicated in the consent form.

Exclusion Criteria

1. Failure to meet any one of the inclusion criteria.
2. Smokers
3. Known history of AIDS, hepatitis, a history or presence of clinically important endocrine conditions (including Type 1 or Type 2 diabetes mellitus), pulmonary, biliary or gastrointestinal (GI) disorders or new onset cardiovascular disease within 6 months of screening (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke).
4. Use of antibiotics within 1 week of screening.
5. Use of probiotic supplements within 1 week of screening.
6. Use of medications known to influence carbohydrate metabolism, GI function or appetite, including, but not limited to adrenergic blockers, diuretics, thiazolidinediones, metformin and systemic corticosteroids within 4 weeks of the screening visit, or with any condition which might, in the opinion of the Investigator, either: a) make participation dangerous to the subject or to others, b) affect the results, or c) influence the ability of the subject to comply with study procedures.
7. Major trauma or surgical event within 3 months of screening.
8. Unwillingness or inability to comply with the experimental procedures and to follow study safety guidelines.
9. Known intolerance, sensitivity or allergy to any ingredients in the investigational agent.
10. Extreme dietary habits, as judged by the Investigator (i.e. Atkins diet, very high protein diets, etc.).
11. History of cancer in the prior two years, except for non-melanoma skin cancer.
12. Recent history (within 12 months of screening) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as > 14 drinks per week (1 drink=12 oz beer, 5 oz wine, or 1.5 oz distilled spirits).
13. Pregnancy or breastfeeding.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-06-22 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Fasting blood lipid levels | Baseline vs. Week 7
  triglycerides, HDL and LDL cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wolever, MD/PhD, Principal Investigator — INQUIS Clinical Research
Locations (1):
- Inquis Clinical Research, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No